CLINICAL TRIAL: NCT04261621
Title: Early Identification of SEPsis SIGNs in Emergency Department
Acronym: SepSIGN
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Collaborators: Vanderbilt University Medical Center (Other); Centre d'Investigation Clinique - Limoges (Unknown)
Responsible Party: Sponsor
Other Study IDs: SepSIGN
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Infection; Sepsis
Keywords: Infection; Sepsis; Worsening; Emergency Department
MeSH Terms: conditions — Infections; Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Four types of samples are taken for the study per patient at T0:
  * Up to 3ml of urine
  * 2.5 mL of whole blood collected in a PAXgene tube
  * 7 mL collected in a dry tube for serum biobank
  * 7 mL collected in a lithium heparin tube for plasma biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective of SepSIGN project is to validate biomarkers able to predict the clinical worsening of patients freshly admitted at Emergency Department. Targeted population is adult patients, freshly admitted at ED, with a suspected or confirmed infection.

DETAILED DESCRIPTION:
Sepsis is an important health issue with considerable socio-economic consequences. In 2017, the World Health Association made sepsis a global health priority, and has adopted a resolution to improve the prevention, diagnosis, and management of sepsis.

Over the last decade, a decrease in the mortality rate has been observed; in particular thanks to improved management, more appropriate intervention approaches in the Emergency Department (ED) and better recognition of organ failure. This statement is based on qSOFA and SOFA scores from the international Sepsis-3 definition. Sepsis-3 can help front-line clinicians detect severe patients with a higher risk of mortality but does not predict the clinical deterioration especially in patients without initial organ dysfunction. Furthermore, studies still demonstrate that 20% of patients with infection or uncomplicated sepsis experience disease worsening within 72 hours after ED admission.

Symptoms and signs of sepsis are variable and this makes clinical recognition and assessment very difficult in particular on Emergency Department (ED) patients due to their infectious illness background and the frequent comorbidities.

Unfortunately, as of today, no biological marker has yet been validated to appropriately predict early deterioration in unselected patients admitted to the ED with acute infection, irrespective of their clinical presentation. Physiology of sepsis is complex and some underlying dysfunction could already exist in the early phase of sepsis before patients meet diagnostic criteria. Thus, patients may be clinically asymptomatic at the origin of organ failure. As a result, doubtful patients are often over-hospitalized while they could be treated at home, leading to overcrowding and extra costs for hospitals In these conditions, the main challenge of ED clinicians is differentiating mild infections from life-threatening ones in the heavy workload of ED environment. Objective of SepSIGN project is to validate biomarkers able to predict the clinical worsening of patients freshly admitted at Emergency Department. Targeted population is adult patients freshly admitted at ED, whom blood samples will serve to validate candidate markers.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria:

* Delay between ED presentation and inclusion must not exceed 12h
* Age 18 years or greater
* Acute infection suspected or confirmed
* That fulfills at least two of the following systemic inflammatory response syndrome (SIRS) criteria:

  * Temperature > 38°C (100.4°F) or < 36°C (96.8°F)
  * Heart rate > 90 bpm
  * Respiratory rate > 20 cycles/min or PaCO2 < 32 mmHg
  * Leukocyte > 12000/mm3 or < 4000/mm3 or 10% bands
* With a delta SOFA < 2 from baseline
* At Risk for deterioration defined as:

  1. any patient that the emergency department physician has admitted or intends to admit as an inpatient* to the hospital.
  2. patients discharged home (outpatient**) who are either i) >65 years old or ii) diagnosed with pneumonia

Exclusion Criteria:

* Unable to obtain a valid and written consent from a patient or their legally authorized representative in accordance with the local regulatory instances (this include in FR: Person not affiliated to a health insurance scheme, or not a beneficiary of such a scheme. Persons who are the subject of a legal protection order. Person with restricted freedom following a legal or administrative decision and a person admitted without their consent pursuant to Articles L.3212-1 and 3213-1, which are not included in Article L.1122-8 of the French Public Health Code.)
* Known pregnancy, in labor or breastfeeding
* Patients with isolated uncomplicated pharyngitis, sinusitis, or otitis media
* Infectious symptoms present for > 5 days prior to presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient freshly admitted to Emergency department
Sampling Method: Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
number of patients with deterioration within 72-hour period following T0 (enrollment) | Up to 72 hours after admission
  clinical deterioration of a patient at any time during the 72-hour period following T0 (enrollment), which is defined as any of the following:
  * increase of SOFA score ≥ 2 points
  * need of new organ support (respiratory, circulatory, renal)
  * death An Endpoint Adjudication Committee (EAC) composed of acute care specialists will apply these criteria. This EAC will also confirm /exclude the presence of infection at T0 (enrollment) based on all information available in eCRF.

SECONDARY OUTCOMES:
Number of Participants that have been re-admission | Up to 28 days after admission
  Re-admission in hospital any time from T0 to T72h (for patients who have been admitted) OR Admission any time from T0 to T72h (for patients who were discharged from the emergency department)
Number of patients with Early and late mortality | Up to 28 days after admission
  Early and late mortality defined by vital status of patients (alive or dead) at Day 28. This information will be collected on the associated eCRF or obtained using follow up procedures (including telephone call) for the patients discharged.
number of patients with confirmed bacterial and viral infection | Up to 28 days after admission
  the adjudication committee will also confirm site of infection and diagnosis of infection A. Confirmed sites of infections B. Infection status (Infection DEFINITELY present / Infection LIKELY present / Infection LIKELY NOT present / NON INFECTIOUS diagnosis identified) C. Viral versus bacterial infections

CONTACTS AND LOCATIONS:
Locations (12):
- United States (4):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington
- France (7):
  - CH Henri Mondor Aurillac, Aurillac
  - CHU Grenoble alpes, La Tronche
  - CHU Dupuytren, Limoges
  - Hopital Edouard Herriot, HCL, Lyon
  - CH de Montauban, Montauban
  - Hôpital Saint-Antoine AP-HP, Paris
  - Hôpital Trousseau CHRU, Tours
- Centre Hospitalier Princesse Grace, Monaco, Monaco